CLINICAL TRIAL: NCT06609304
Title: Prospective Clinical Study of Axicabtagene Ciloleucel for Consolidation After First-line Treatment of High-risk Large B-cell Lymphoma
Brief Title: Axicabtagene Ciloleucel for Consolidation After First-line Treatment of High-risk Large B-cell Lymphoma
Acronym: axi-cel
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, Professor, Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA2024-252
Record Dates: First submitted 2024-08-28; First posted 2024-09-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- axi-cel treatment (Experimental)
  Interventions: Biological: Axicabtagene Ciloleucel

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — Axicabtagene Ciloleucel at 2.0×10^6/Kg

SUMMARY:
The goal of this clinical trial is to learn if Axicabtagene Ciloleucel (axi-cel) works for consolidation after first-line treatment of high-risk Large B-cell Lymphoma (LBCL). It will also learn about the safety of axi-cel treatment. The main questions it aims to answer are:

* Does axi-cel treatment result in prolonged clinical benefit to patients with high-risk LBCL after first-line treatment?
* What medical problems do participants have when receiving axi-cel treatment?

In this investigator-initiated, single-arm clinical trial, participants will:

* Receive atezolizumab treatment at 2.0×10^6 cells/Kg as a one-time therapy.
* Visit the clinic as instructed for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form;
2. 18-70 years of age (inclusive);
3. Previously untreated CD19-positive large B-cell lymphoma;
4. Anticipated survival ≥12 weeks;
5. Adequate bone marrow reserve prior to apheresis
6. Appropriate organ function:
7. Eastern Cooperative Oncology Group (ECOG) Physical Status Score of 0 or 1; 8. Absence of CNS lymphoma;

9. Negative blood/urine pregnancy test in women of childbearing age.

Exclusion Criteria:

1. History of allergy to any of the components of the cell product;
2. History of stem cell transplantation;
3. History of organ transplantation;
4. Presence of active infections;
5. Current or history of central nervous system disorders;
6. Previous treatment with other modified T-cell therapy;
7. Previous treatment with anti-CD19/CD3 or other anti-CD19 therapies;
8. Malignancies other than those indicated for this trial;
9. History of any prior systemic immune checkpoint therapy;
10. History of short-acting cell growth factors or haematopoietic agonists/stimulants ;
11. History of a live vaccine within 3 months prior to screening;.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
one year PFS | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Department of Oncology, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No